CLINICAL TRIAL: NCT04724616
Title: CARTOON: CoronAviRus educaTional prOgram fOr childreN to Promote Knowledge and Hygiene Measures and Dispel Fear During the COVID- 19 Pandemic
Brief Title: CARTOON: CoronAviRus (COVID-19) educaTional prOgram fOr childreN
Acronym: CARTOON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Philipp Steinbauer, Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2128/2020
Record Dates: First submitted 2021-01-10; First posted 2021-01-26 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Covid19; Pediatric Psychiatric Disorder; Psychological Stress
Keywords: Educational Program; education
MeSH Terms: conditions — COVID-19; Neurodevelopmental Disorders; Stress, Psychological | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants received no specific educational program
- Intervention Group (Experimental): Participants received our educational program for five days, with one teaching session per day. Every teaching session will be conducted for 60 minutes in a group of up to 6 children by a trained member of our staff.
  Interventions: Other: Educational Program (CARTOON)

INTERVENTIONS:
Other: Educational Program (CARTOON) — CARTOON is an interdisciplinary psychoeducational intervention program. It consists of five teaching sessions: 1) hand hygiene, not grasping the face, 2) sneezing etiquette, 3) wearing a mask, 4) social distancing, and 5) theoretical knowledge about the coronavirus. Using special exercises and games, information about the coronavirus is conveyed in a child friendly manner.
  Other Names: Education; Psycho-educational intervention
  Arms: Intervention Group

SUMMARY:
Our study aims to investigate whether our CoronAviRus educaTional prOgram fOr children (CARTOON) facilitates the adherence to hygiene measures and is feasible to dispel fear in preschool children (3-6 years old) during the pandemic.

DETAILED DESCRIPTION:
This prospective randomized controlled trial will be performed at four kindergartens in Vienna, Austria. About 60 children between three and six years of age attending kindergarten will be included in the study. Prior inclusion in the study eligible adults have to sign a parental consent form. We will randomly assign 30 children to the intervention group (n=30) and 30 children to the control group (n=30). Depending on the randomization (intervention group vs. control group), children either receive our CARTOON (intervention group) or no educational training (control group).

ELIGIBILITY:
Inclusion Criteria:

* Children between three and six years who are attending kindergarten
* consent of the parents and the participants

Exclusion Criteria:

* physically unable to complete any of the training exercises
* German skills not good enough to follow the instructions

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Change of Emotional Outcome | Baseline (before the intervention), 1 day after the intervention and three months after the intervention
  For the assessment of emotional wellbeing, fear, and burden during the pandemic we will use the emotional scale which measure feelings including emotional wellbeing, fear, and burden.
  Since it is often hard for children to describe their own feelings with words, we will use the emotional scales of Gräßler and colleagues. These scales use child-friendly illustrated pictures and can be used to support the children in naming their feelings including emotional wellbeing, fear, and burden.
Change of Knowledge Outcome | Baseline (before the intervention), 1 day after the intervention and three months after the intervention
  The corona quiz consists of a 18-item questionnaire and covers theoretical and practical knowledge. Content validity of the knowledge test was reviewed by an expert panel consisting of three psychologists with expertise in children health, one kindergarten teacher, and one pediatrician.
Baseline Behavior of the Participants | Baseline (before the intervention)
  Behavior will be assessed by using the parent and teacher reported Child Behavior Checklist (CBCL). The CBCL is a questionnaire for parents and teachers revealing behavioral problems of children and adolescents. In the CBCL/1.5-5, two evaluation methods are available. In the first evaluation method, questions are grouped in seven empirically based problem scales including emotionally reactive, anxious/depressed, aggressive behavior, attention problems, somatic complaints, sleep problems, and withdrawn.

SECONDARY OUTCOMES:
Nationality of parents | Baseline (before the intervention)
  Is there a correlation of the Nationality of the parents with emotional and knowledge outcomes of the children
First language of parents | Baseline (before the intervention)
  Is there a correlation of the first language of the parents with emotional and knowledge outcomes of the children
Highest degree of school education | Baseline (before the intervention)
  Is there a correlation of the highest degree of school education of the parents with emotional and knowledge outcomes of the children
Profession of the parents | Baseline (before the intervention)
  Is there a correlation of the profession of the parents with emotional and knowledge outcomes of the children
Financial standing of the parents | Baseline (before the intervention)
  Is there a correlation of the financial standing of the parents with emotional and knowledge outcomes of the children
Housing conditions of the family | Baseline (before the intervention)
  Is there a correlation of the housing condition of the family with emotional and knowledge outcomes of the children
Psychological or physical illness in the family | Baseline (before the intervention)
  Is there a correlation of the psychological or physical burden in the family with emotional and knowledge outcomes of the children

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Steinbauer, Dr., Principal Investigator — Comprehensive Center For Pediatrics, Division of Neonatology, Intensive Care Medicine and Neuropediatrics
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Steinbauer P, Bichler M, Fuiko R, Seferagic S, Haas H, Lisy T, Weinmuller S, Berger A, Olischar M, Panagl A, Giordano V. CARTOON-based educational intervention for children to foster hygiene knowledge and emotional resilience in preschool children: a randomized controlled trial. Front Pediatr. 2025 Apr 11;13:1514793. doi: 10.3389/fped.2025.1514793. eCollection 2025. PMID 40292121